CLINICAL TRIAL: NCT05682846
Title: Impact of Serum Phosphorus Level Optimization on Weaning From Mechanical Ventilation in Adult ICU Patients
Brief Title: Optimization of Serum Phosphorus Level and Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Mahmoud Abdelghany, Master's student in Clinical Pharmacy and Pharmacy Practice, Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0107114
Record Dates: First submitted 2022-12-07; First posted 2023-01-12 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Mechanical Ventilation
Keywords: Mechanical ventilation; Phosphorus; Critical illness; Ventilator weaning
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (Experimental): Optimization of serum phosphorus to ≥ 3.5 and ≤ 4.5 mg/dL (Average 4mg/dL) using Sodium glycerophosphate pentahydrate solution.
  Sodium glycerophosphate pentahydrate 20ml solution (20 mmol glycerophosphate) dose will be given once daily till the target serum phosphorus level is achieved.
  Interventions: Drug: Sodium glycerophosphate pentahydrate solution
- Control group (No Intervention): Maintaining serum phosphorus level at ≥ 2.5 and < 3.5 mg/dL.

INTERVENTIONS:
Drug: Sodium glycerophosphate pentahydrate solution — Glycophos is a 20 ml vial of Sodium glycerophosphate pentahydrate containing 1 mmol glycerophosphate and 2 mmol sodium per ml
  Other Names: Glycophos
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to test the impact of serum phosphorus level optimization on weaning from mechanical ventilation in adult ICU patients in Alexandria University Hospitals.

The main questions it aims to answer are:

* Does serum phosphorus level optimization affect the duration of mechanical ventilation?
* Is serum phosphorus level optimization associated with successful weaning from mechanical ventilation?

In critically ill patients, phosphorus supplementation is done using Sodium glycerophosphate pentahydrate solution.

DETAILED DESCRIPTION:
Investigators will document patients' data in terms of independent variables and will randomly allocate the participants into one of the two study groups mentioned below.

* Control group, defined by maintaining serum phosphorus level at ≥ 2.5 and < 3.5 mg/dL.
* Intervention group, defined by optimization of serum phosphorus P to ≥ 3.5 and ≤ 4.5 mg/dL (Average 4mg/dL).

Regression and comparative statistics will be used to determine whether the optimum serum phosphorus level offers a benefit in terms of the duration of mechanical ventilation and the success of weaning from mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult mechanically ventilated ICU patients.
* Age ≥ 18 years.

Exclusion Criteria:

* Age <18 years
* Hypernatremia
* Permanent or prolonged mechanical ventilation
* Hyperphosphatemia which might occur in the following conditions:
* Chronic kidney disease and end stage renal disease
* Parathyroid disorders
* Cancer patients at risk of tumor lysis syndrome
* Immobility
* Body weight < 50 Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The duration of mechanical ventilation. | 4 months
  Comparison of mechanical ventilation days for patients in the two study groups.
Weaning from mechanical ventilation. | 4 months
  Association of serum phosphorus level optimization to ≥ 3.5 and ≤ 4.5 mg/dL with success of weaning from mechanical ventilation.

SECONDARY OUTCOMES:
Length of ICU stay | 4 months
  Change in the ICU length of stay in the intervention group with respect to the control group
ICU mortality | 4 months
  Change in the ICU mortality in the intervention group with respect to the control group.
Cost effectiveness analysis | 4 months
  Cost-effectiveness analysis of serum phosphorus level optimization.

CONTACTS AND LOCATIONS:
Overall Officials: Magda A El-Massik, PhD, Principal Investigator — Professor of Pharmaceutics, Alexandria University; Haitham M Tammam, PhD, Principal Investigator — Associate professor of Critical Care Medicine, Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Assistant Professor of Clinical Pharmacy, Alexandria University; Marawan M ElBourini, PhD, Principal Investigator — Lecturer in Critical Care Medicine, Alexandria University; Yasmin M Abd Elghany, PharmD, Principal Investigator — Master's student in Clinical Pharmacy and Pharmacy Practice, Alexandria University.
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aubier M, Murciano D, Lecocguic Y, Viires N, Jacquens Y, Squara P, Pariente R. Effect of hypophosphatemia on diaphragmatic contractility in patients with acute respiratory failure. N Engl J Med. 1985 Aug 15;313(7):420-4. doi: 10.1056/NEJM198508153130705. PMID 3860734
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Liu B, Cheng Y, Shen F, Wang Y, Wu Y, Yao L, Liu Y, Gou X. [Hypophosphatemia is associated with poor prognosis of critically ill patients: a meta-analysis of 1 555 patients]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2018 Jan;30(1):34-40. doi: 10.3760/cma.j.issn.2095-4352.2018.01.007. Chinese. PMID 29308755
- [Background] Sin JCK, King L, Ballard E, Llewellyn S, Laupland KB, Tabah A. Hypophosphatemia and Outcomes in ICU: A Systematic Review and Meta-Analysis. J Intensive Care Med. 2021 Sep;36(9):1025-1035. doi: 10.1177/0885066620940274. Epub 2020 Aug 12. PMID 32783487
- [Background] Padelli M, Leven C, Sakka M, Plee-Gautier E, Carre JL. [Causes, consequences and treatment of hypophosphatemia: A systematic review]. Presse Med. 2017 Nov;46(11):987-999. doi: 10.1016/j.lpm.2017.09.002. Epub 2017 Oct 28. French. PMID 29089216
- [Background] Sahetya S, Allgood S, Gay PC, Lechtzin N. Long-Term Mechanical Ventilation. Clin Chest Med. 2016 Dec;37(4):753-763. doi: 10.1016/j.ccm.2016.07.014. Epub 2016 Oct 14. PMID 27842754
- [Background] Santibanez-Velazquez M, Medina-Garcia G, Ocharan-Hernandez ME. Association of independent risk factors with post-extubation failure in patients undergoing mechanical ventilation weaning. Gac Med Mex. 2020;156(6):539-545. doi: 10.24875/GMM.M21000493. PMID 33877109
- [Background] Wang L, Xiao C, Chen L, Zhang X, Kou Q. Impact of hypophosphatemia on outcome of patients in intensive care unit: a retrospective cohort study. BMC Anesthesiol. 2019 May 24;19(1):86. doi: 10.1186/s12871-019-0746-2. PMID 31122196
- [Background] Wozniak H, Dos Santos Rocha A, Beckmann TS, Larpin C, Buetti N, Quintard H, Pugin J, Heidegger CP. Hypophosphatemia on ICU Admission Is Associated with an Increased Length of Stay in the ICU and Time under Mechanical Ventilation. J Clin Med. 2022 Jan 24;11(3):581. doi: 10.3390/jcm11030581. PMID 35160032